CLINICAL TRIAL: NCT00020540
Title: Treatment Of Patients With Metastatic Melanoma And Renal Cancer With A Combination Of Flt3L And CD40L
Brief Title: Biological Therapy in Treating Patients With Metastatic Melanoma or Metastatic Kidney Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000068601; NCI-01-C-0121; NCI-1035; NCT00012532 (obsolete NCT alias)
Record Dates: First submitted 2001-07-11; First posted 2004-04-05 (Estimated); Last update posted 2015-04-30 (Estimated); Status verified 2002-04

CONDITIONS: Kidney Cancer; Melanoma (Skin)
Keywords: stage IV renal cell cancer; recurrent renal cell cancer; stage IV melanoma; recurrent melanoma
MeSH Terms: conditions — Kidney Neoplasms; Melanoma; Carcinoma, Renal Cell | interventions — CD40 Ligand; flt3 ligand protein

INTERVENTIONS:
Biological: recombinant CD40-ligand
Biological: recombinant flt3 ligand

SUMMARY:
RATIONALE: Biological therapies such as flt3L and CD40-ligand use different ways to stimulate the immune system and stop cancer cells from growing. Biological therapy may be an effective treatment for metastatic melanoma and metastatic kidney cancer.

PURPOSE: Phase I trial to study the effectiveness of flt3L combined with CD40-ligand in treating patients who have metastatic melanoma or metastatic kidney cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the maximum tolerated dose of CD40-ligand when combined with fixed-dose flt3 ligand in patients with metastatic melanoma or renal cell cancer.

OUTLINE: This is a dose-escalation study of CD40-ligand. Patients receive fixed-dose flt3 ligand subcutaneously (SC) daily on days 1-14 and CD40-ligand SC daily on days 12-16. Treatment continues every 28 days for a maximum of 6 courses in the absence of unacceptable toxicity or disease progression. Cohorts of 3 to 6 patients receive escalating doses of CD40-ligand until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 6 patients experience dose-limiting toxicity. Patients with progressive disease after 2 courses may be eligible to receive high-dose interleukin-2 (IL-2) standard therapy.

PROJECTED ACCRUAL: A total of 5 patients were accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed metastatic renal cell cancer or melanoma Measurable disease

PATIENT CHARACTERISTICS: Age: 16 and over Performance status: ECOG 0-1 Life expectancy: More than 3 months Hematopoietic: WBC at least 3,000/mm3 Platelet count at least 90,000/mm3 No coagulation disorders Hepatic: Bilirubin no greater than 1.6 mg/dL AST and ALT less than 2.5 times normal Hepatitis B surface antigen negative Renal: Creatinine no greater than 2.0 mg/dL Cardiovascular: No major active medical illness of the cardiovascular system (e.g., cardiac ischemia, myocardial infarction, or cardiac arrhythmia) Pulmonary: No major active medical illness of the respiratory system (e.g., obstructive or restrictive pulmonary disease) Other: Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception No active systemic infections No history of autoimmune disorders HIV negative

PRIOR CONCURRENT THERAPY: Biologic therapy: At least 3 weeks since prior biologic therapy No prior systemic flt3 ligand or CD40-ligand Chemotherapy: At least 3 weeks since prior chemotherapy Endocrine therapy: At least 3 weeks since prior endocrine therapy No concurrent systemic steroids Radiotherapy: Prior localized radiotherapy for renal cell cancer or melanoma allowed Surgery: Prior surgery for renal cell cancer or melanoma allowed

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2001-03

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Hwu, MD, Study Chair — NCI - Surgery Branch
Locations (1):
- Surgery Branch, Bethesda, Maryland, United States